CLINICAL TRIAL: NCT02134444
Title: Comparison of Clinical and Game-based Rehabilitation for Balance Impairments and Gaze Dysfunction in Clients With Vestibular Disorders
Brief Title: Game Based Vestibular Exercise for Home Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: not yet conducted
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2014-04

CONDITIONS: Peripheral Vestibular Disorders; Dizziness
Keywords: Dizziness; Vertigo; Vestibular Diseases; Vestibular Neuritis; Labyrinth Diseases; Ear Diseases; Vestibular rehabilitation; Telerehabilitation; Gaze control; Balance
MeSH Terms: conditions — Dizziness; Vertigo; Vestibular Diseases; Vestibular Neuronitis; Labyrinth Diseases; Ear Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Experimental group will receive the assigned intervention which is a game-based rehabilitation program delivered at home.
  Interventions: Behavioral: Experimental group
- Control group (Active Comparator): Control group will receive a vestibular rehabilitation program which will include the Herdman gaze stabilization exercises and balance training program.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Experimental group — Experimental group will receive a game-based exercise program delivered at home. This includes provision of a head-mounted motion mouse. This provides a treatment tool applied to gaze control, and allows incorporation of balance exercises. It also allows many different therapeutic exercises to be coupled to a wide range of inexpensive commercial computer games. Participants will attend 3 clinical sessions during which time the home therapy programs will be established and training in the use of the motion mouse and games will be provided. The treating physiotherapist will attend the participant's home to ensure proper set-up and operation of the computer applications. Participants will be asked to perform their respective home programs four times per week for 20 minutes per session.
  Arms: Experimental Group
Behavioral: Control group — Control group will receive a vestibular exercise program which will include the Herdman gaze stabilization exercises and balance training program. This program is presently a standard of vestibular care. Participants will attend an out-patient physical therapy clinic once a week for 12 weeks. The program also includes a 20 minute home exercise program prescribed 4 times per week.
  Arms: Control group

SUMMARY:
Study Description and Purpose:

The vestibular sense organs of the inner ear consist of the semi-circular canals and otolith end organs. These organs contain specialized gravito-inertial sensors that sense angular and linear head acceleration. The input from these sensors is required to stabilize gaze position during head motion, and provide an absolute frame of reference with respect to gravity, thus providing a vertical spatial reference for body orientation and balance. Disease or damage of the vestibular sense organs causes a range of distressing symptoms and functional problems for people that could include loss of balance, gaze instability, disorientation and dizziness. A novel computer based rehabilitation system with therapeutic gaming application has been developed. This method allows different gaze and head movement exercises to be coupled to a wide range of inexpensive, commercial computer games. It can be used in standing and thus graded balance demands using a sponge pad can be incorporated into the program.

Study Objective:

1. Test the therapeutic effectiveness of the TRP delivered in the home compared to usual care delivered in an out-patient physical therapy clinic on measures of balance (standing and walking) , gaze control, dizziness, and health related quality of life in individuals with peripheral vestibular disorders.
2. Compare trajectory of change in electronic gaze performance measures obtained during each therapy session of each participant assigned to the home Telerehabilitation.

Hypothesis:

Investigators believe the Telerehabilitation platform to be a cost-effective delivery of rehabilitation. Additionally motivation to perform tedious home programs can be improved with engaging, fun and interactive computer gaming as part of the rehabilitation process. It is hypothesized the home game-based Telerehabilitation program will result in greater improvements in dynamic balance control, gaze control, and dizziness, in individuals with peripheral vestibular disorders as compared to a typical out-patient physical therapy regimen.

DETAILED DESCRIPTION:
Protocol

Design & Methodology:

This study will adopt a randomized clinical trial design. Recruitment and screening (including diagnostics) will be coordinated by co-applicant, Dr. Jordon Hochman, department of Otolaryngology, Karen Reimer, and Andrea Giacobbo,; Physical Therapists.

Inclusion criteria:

Consist of (a) age 18 to 65 , (b) diagnosed with unilateral peripheral vestibular hypo function based on a detailed neuro-otological and neuro-orthoptic analysis to include binocular electro-oculography with caloric testing, and (c) have a home computer running Windows or Mac OS.

Exclusion criteria:

Consist of those with CNS disorders for example CVA, Multiple Sclerosis, epilepsy, migraines, concussion recent fractures of the lower extremities or vertebra, advanced hip/knee OA , and cardiac disease. Participants will be randomly assigned to either the Control group (active comparator) or Experimental group (therapeutic gaming). Participants will be blinded to the treatment. The treating therapist will know who is receiving the home or out-patient clinical program.

Control group will receive; (a) Herdman gaze stabilization exercises, (b) optokinetic exercises, and (c) balance exercises using sponge pads. These exercises are presently a standard of vestibular care. Participants will attend an out-patient physical therapy clinic once a week for 8-10 weeks. The program also includes a 20 minute home exercise program prescribed four times per week.

Experimental group: Will receive the game-based rehabilitation program delivered at home. The program for gaze will include provision of the motion mouse (Gyration). This approach provides a highly flexible treatment tool applied to train gaze control, and allows incorporation of graded balance demands. The use of this HID compliant computer input device allows many different therapeutic exercises to be coupled to a wide range of inexpensive commercial computer games. Though initially designed for clinical use, with the easy to use and inexpensive motion sense mouse and computer games this intervention approach can be extended to home settings. Many therapeutic exercises and activities (singly or in combination) can be used to practice a variety of gaze and balance skills, and, importantly, while playing fun computer games.

Participants will attend three clinical sessions during which time the home therapy programs will be established and training in the use of the computer, motion mouse and games will be provided. Based on clinical experience and pilot data, three sessions is sufficient before initiating the home program.16 The treating physiotherapist will attend the participant's home to ensure proper set-up and operation of the TRP equipment and computer applications. Participants will be asked to perform their respective home programs four times per week for 20 minutes per session. They will receive a phone call at one week to assess their ability to manage their home program. Thereafter participants will attend for clinical follow-up once per month.

Recording and Data Analysis The following information will be collected at baseline prior to start of the interventions; age, gender, work history, occupation and (history of disease/injury process, and current medications. Assessor will be blinded to participant assignments.

Primary Outcome Measures:

1. Clinical Test of Sensory Interaction in Balance (CTSIB); performance-based measure of balance under altered sensory conditions).
2. Dizziness Handicap Inventory (DHI), is a self-rating questionnaire based on 25 questions used to quantify a client's perception of his or her dizziness and its impact on their life.

Secondary outcome measures:

1. Computerized Visual tracking test (CVT), involves tracking a bright visual target moving horizontally left and right on a computer display in a sinusoidal fashion for several cycles, and at predetermined speeds. The application records (80 Hz) coordinates of both reference and head cursors. Coefficient of determination (COD) will be computed based on total and average residual difference between trajectories of the reference and head cursor motions. A value approaching one equates to excellent gaze performance. This test will be performed in standing and while walking on a treadmill at 0.9 m/s.
2. Participants in the experimental group will be given the visual tracking game application for home use. The game software automatically logs reference and head cursor coordinates (gaze performance) during the visual tracking task and saves the data to a coded and time stamped computer file (anatomized). Participants will be asked to play the tracking task (in standing at the beginning of every training session. This will involve three short tests of 45 seconds at three tracking speeds. The application automatically saves the logged data file, and the clients can either e-mail the files to the investigator, or save on a flash drive provided and return at a follow-up visit.
3. Spatiotemporal gait variables and walking stability measures. This is included to examine whether the exercise program transfers to walking. A treadmill instrumented with a pressure mat (Vista Medical, CA) will be used to record vertical foot forces for each step during walking trials of 1 minute at 0.9 m/s, and thus data for 40 consecutive steps.
4. Participants will be ask to complete a log of dates and duration of each exercise session, and submit either a paper version or by e-mail.

Statistical Analysis & Power Assessment: Descriptive statistics, including means, standard deviations, frequencies, and percentages, will be used to describe the experimental and control groups on the baseline demographic variables. Differences between the groups on the outcomes will be tested using t-tests and tests of independence.

To achieve Objective 1, we will test the difference between experimental and control groups on continuous and normally distributed outcome measures using analysis of covariance, with the dependent variable being the post-intervention measurement of the outcome, the covariate being the pre-intervention measurement, and group membership as the between-subjects effect. Descriptive statistics, including measures of skewness and kurtosis, will be used to assess departures from the assumptions of a normal distribution of responses. If the distribution contains extreme observations, a robust ANCOVA statistic will be adopted. To test differences between experimental and control groups on discrete outcomes, such as counts of number of times participants feel dizzy during their daily activities, we will use a Poisson regression model, with the dependent variable being a count of the number of relevant events, the covariate being the pre-intervention measurement, and group membership as the between-subjects effect.

To analyze the longitudinal data associated with Objective 2, we will use a mixed-effects regression model with time as the random effect and group as the fixed effect. This model will be adopted because it accounts for clustering of repeated measurements within study participants and uses all available longitudinal data (i.e., it does not result in case-wise deletion of study participants due to missing observations.

Based on pilot data for the primary outcome (i.e., CTSIB), we conducted a power analysis of the required sample size to test the difference between the experimental and controls groups at the post-intervention measurement occasion (i.e., objective 1). The pilot data showed a standardized effect size of 0.80. Assuming the number of model covariates to be 3, the proportion of variance explained by these covariates to be 10%, and a two-tailed test of the null hypothesis of no group difference at p = .05, a sample size of 46 is required. We expect an attrition rate of 20% over the study observation period for objective 2. Given this, we propose to recruit a sample of N = 56 individuals to participate, with equal numbers to be recruited to the treatment and control groups.

ELIGIBILITY:
Inclusion criteria:

1. Age between 20-60
2. English speaking
3. Diagnosed with unilateral or bilateral peripheral vestibular hypo function based on a detailed neuro-otological and neuro-orthoptic analysis to include binocular electro-oculography with caloric testing;
4. Have a home computer running Windows or Mac OS. 5 Adequate hearing and vision acuity

Exclusion Criteria:

1. Those with CNS disorders for example CVA, Multiple Sclerosis, epilepsy, migraines.
2. Recent fractures of the lower extremities or vertebra, advanced hip/knee OA ,
3. Cardiac disease .

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Standing Balance | Pre and post intervention of 12 weeks
  This will be measured by performing a) Clinical Test of Sensory Integration of Balance and b) Five - Time Sit-to-Stand Test.
  Centre of Foot Pressure (COP) is recorded during test conditions and root mean square (RMS) and total Path Length ) in Medial-Lateral and Anterior-Posterior Directions is quantified.
Dizziness Handicap Inventory (DHI) | Pre and post intervention of 12 weeks
  It is a self-rating questionnaire based on 25 questions used to quantify a client's perception of his or her dizziness and its impact on their life.
Computerized Visual Tracking Performance | Pre and post intervention of 12 weeks
  A computer application has been developed which involves tracking a bright visual target moving horizontally left and right on a computer display in a sinusoidal fashion for several cycles, and at predetermined speeds. This procedure requires vestibular function and smooth pursuit to coordinate eye and head motions during the active head tracking task. The computer application records (80 Hz) coordinates of both reference and head cursors. Coefficient of determination (COD) will be computed based on total and average residual difference between trajectories of the reference and head cursor motions. A value approaching one equates to excellent gaze performance. This test will be performed in sitting, standing and while walking on a treadmill at 0.9 m/s
Spatial - temporal gait variables during treadmill walking with and without visual tracking task. | Pre and post intervention of 12 weeks
  It will be measured by asking the participants to walk on a treadmill for 1 minute which is instrumented with a pressure mat at a speed of 0.9 m/s. Average and coefficient of variation will be obtained for the following parameters: swing time, step time, step length and step width.
  Participants will repeat the:
  1. Baseline walk not engaged in any visual tracking or head movement task
  2. While performing the CDVA visual tracking task described above for 45 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, PT, PhD, Principal Investigator — University of Manitoba; Jordan Hochman, MD, Principal Investigator — University of Manitoba; Lisa Lix, PhD, Principal Investigator — University of Manitoba; Christine Wu, Principal Investigator — University of Manitoba; Karen Reimer, PT, M.Sc., Principal Investigator — Private Practice Clinician; Andrea Giacobbo, PT, Principal Investigator — Private Practice Clinician
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Szturm T, Betker AL, Moussavi Z, Desai A, Goodman V. Effects of an interactive computer game exercise regimen on balance impairment in frail community-dwelling older adults: a randomized controlled trial. Phys Ther. 2011 Oct;91(10):1449-62. doi: 10.2522/ptj.20090205. Epub 2011 Jul 28. PMID 21799138
- [Background] Desai A, Goodman V, Kapadia N, Shay BL, Szturm T. Relationship between dynamic balance measures and functional performance in community-dwelling elderly people. Phys Ther. 2010 May;90(5):748-60. doi: 10.2522/ptj.20090100. Epub 2010 Mar 11. PMID 20223944
- [Background] Szturm T, Maharjan P, Marotta JJ, Shay B, Shrestha S, Sakhalkar V. The interacting effect of cognitive and motor task demands on performance of gait, balance and cognition in young adults. Gait Posture. 2013 Sep;38(4):596-602. doi: 10.1016/j.gaitpost.2013.02.004. Epub 2013 Mar 9. PMID 23477841
- [Background] Szturm T, Wu c. etal. (2013). Technology-assisted & motivational program for a blended approach to manage balance gaze mobility and cognitive decline with age. OA Evidence-Based Med. Apr;1):1.
- [Background] Lockery D, Peters JF, Ramanna S, Shay BL, Szturm T. Store-and-feedforward adaptive gaming system for hand-finger motion tracking in telerehabilitation. IEEE Trans Inf Technol Biomed. 2011 May;15(3):467-73. doi: 10.1109/TITB.2011.2125976. PMID 21536526
- [Derived] Szturm T, Hochman J, Wu C, Lisa L, Reimer K, Wonneck B, Giacobbo A. Games and Telerehabilitation for Balance Impairments and Gaze Dysfunction: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2015 Oct 21;4(4):e118. doi: 10.2196/resprot.4743. PMID 26490109